CLINICAL TRIAL: NCT03653884
Title: Intra-abdominal Umbilical Vein Aneurysm
Acronym: AVO
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD0716
Record Dates: First submitted 2018-08-24; First posted 2018-08-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-09

CONDITIONS: Obstetric Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnancy with fetal intra-abdominal umbilical vein.: All women with a pregnancy with a partially intra-abdominal umbilical vein aneurysm isolated or associated with other abnormalities découvert lors d'une ultrasonic monitoring.
  Interventions: Diagnostic Test: Ultrasound monitoring

INTERVENTIONS:
Diagnostic Test: Ultrasound monitoring — Ultrasound monitoring is recommended during the third trimester in search of an increase in dilation and especially the appearance of a thrombus. A particular clinical form, related to abnormal umbilical vein involvement in the infra-hepatic portal system, must be individualized because of a high risk of thrombosis. It justifies the realization of an abdominal ultrasound in the first days of life. This is an aneurysm of the umbilical vein when the umbilical vein has a diameter greater than 9 mm, or a diameter of the subhepatic segment of the umbilical vein greater than 50% of the diameter of its intrahepatic segment.

SUMMARY:
The purpose of this study is to investigate the ultrasound characteristics and outcome of pregnancies with fetal Intra-abdominal umbilical vein aneurysm.

DETAILED DESCRIPTION:
Intra-abdominal umbilical vein aneurysm is a rare pathology of the fetal venous system. Its incidence is low, evaluated between 0.4 and 1.1 / 1000.

Intra-abdominal umbilical vein aneurysm is identified as an oval or rounded, anechoic mass located between the abdominal wall and the lower edge of the liver.

It is defined by two criteria: either a diameter greater than 9 mm or a diameter of the subhepatic segment of the umbilical vein greater than 50% of the diameter of its intrahepatic segment.

The complications that can occur during pregnancy are mainly represented by the MFIU, the occurrence of thrombosis and intrauterine growth retardation (IUGR). Their overall frequency is evaluated at 10%.

A complete fetal morphological assessment is necessary to eliminate the presence of other lesions. However, ultrasound monitoring is recommended during the third trimester in search of an increase in dilation and especially the appearance of a thrombus. A particular clinical form, related to abnormal umbilical vein involvement in the infra-hepatic portal system, must be individualized because of a high risk of thrombosis. It justifies the realization of an abdominal ultrasound in the first days of life

ELIGIBILITY:
Inclusion Criteria:

* All patients who have AVO partially intra-abdominal isolated or associated with other abnormalities.
* Patients over the age of 18 who agree to participate in the study after oral information given by the sonographer.
* Any patient seen in 1st intention or 2nd intention.
* Gestational age between 20 and 35 weeks

Exclusion Criteria:

* Patient refusing to participate in the study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients who have AVO partially intra-abdominal isolated or associated with other abnormalities.
  Patients over the age of 18 who agree to participate in the study after oral information given by the sonographer.
  Any patient seen in 1st intention or 2nd intention. Gestational age between 20 and 35 weeks
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
Vital status at birth. | Through study completion, an average of 2 years.
  From birth, it is necessary to evaluate the state of the child. This evaluation is done by the APGAR coefficient. The following actions are systematically performed: place the child on a heating table, aspire mouth, pharynx, nostrils. Specify rapidly, heart and respiratory rhythms, quality of cry, baby's color and responses to skin stimulation. These five criteria rated from zero to two make it possible to determine the Apgar score: it is practiced at one, three, five and ten minutes of life. This assessment helps to guide the behavior of the newborn: if the score is greater than eight to one minute, it means that the newborn has a good adaptation to the ectopic life. If it is less than three to one minute, the newborn is in a state of apparent death involving emergency resuscitation. An intermediate figure, witnessing hypoxia-anoxia, justifies management adapted.

SECONDARY OUTCOMES:
Collection of congenital anomalies and pregnancy Pathologies. | From the inclusion of the patient until the end of pregnancy.
  The complications that may occur during pregnancy are mainly an MFIU, the occurrence of thrombosis and intrauterine growth retardation (IUGR). A complete fetal morphological assessment is necessary to eliminate the presence of other lesions. However, ultrasound monitoring is recommended during the third trimester in search of an increase in dilation and especially the appearance of a thrombus. A particular clinical form, related to abnormal umbilical vein nicking in the infra-hepatic portal system, must be individualized because of a high risk of thrombosis. It justifies the realization of an abdominal ultrasound in the first days of life.
Characteristics of the umbilical vein aneurysm. | From the inclusion of the patient until the end of pregnancy.
  It is defined by two criteria: either a diameter greater than 9 mm, or a diameter of the subhepatic segment of the umbilical vein greater than 50% of the diameter of its intrahepatic segment. There are two forms: an isolated form and a form with other associated abnormalities, which accounts for 29-35% of cases (cardiovascular anomalies, urogenital and hydramnios). Chromosomal abnormalities are found in 6% of cases (T21, T18, T9, triploidy (28% for associated forms and 2% for isolated forms).

CONTACTS AND LOCATIONS:
Overall Officials: Georges MARKOU, Principal Investigator — Hôpital NOVO
Locations (1):
- Centre Hospitalier René-DUBOS, Cergy-Pontoise, France, France